CLINICAL TRIAL: NCT05762471
Title: A Phase 1b/2a, Randomized, Double-blind, Placebo-controlled, Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Doses of GSBR-1290 in Adult Overweight or Obese Healthy Subjects and in Subjects With Type 2 Diabetes Mellitus on Metformin
Brief Title: Phase 1b/2a Study of GSBR-1290 in Adult Overweight or Obese Healthy Subjects and Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gasherbrum Bio, Inc., a wholly owned subsidiary of Structure Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GSBR-1290-02
Record Dates: First submitted 2023-01-25; First posted 2023-03-09 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Overweight or Obesity; Type2 Diabetes Mellitus
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blind study in which the GSBR-1290 and the matching placebo are matching in appearance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Patients will receive once daily doses of study drug (GSBR-1290 or Placebo) for a total of 4 weeks
  Interventions: Drug: GSBR-1290; Drug: Placebo
- Cohort 2 (Experimental): Patients will receive once daily doses of study drug (GSBR-1290 or Placebo) for a total of 4 weeks
  Interventions: Drug: GSBR-1290; Drug: Placebo
- Cohort 3 (Experimental): Patients will receive once daily doses of study drug (GSBR-1290 or Placebo) for a total of 4 weeks
  Interventions: Drug: GSBR-1290; Drug: Placebo
- Cohort 4 (Experimental): HOV participants (Cohort 4) will receive multiple-ascending doses of GSBR-1290 or placebo for a total of 12 weeks
  Interventions: Drug: GSBR-1290; Drug: Placebo
- Cohort 5 (Experimental): Participants with T2DM(Cohort 5) will be randomized to placebo, low-dose, or high-dose arms. Participants in the low-dose, high-dose or placebo arms will receive multiple-ascending doses for 12 weeks
  Interventions: Drug: GSBR-1290; Drug: Placebo

INTERVENTIONS:
Drug: GSBR-1290 — Patients will receive GSBR-1290 or matching Placebo
Drug: Placebo — Patients will receive GSBR-1290 or matching Placebo

SUMMARY:
This study will evaluate safety, tolerability, pharmacokinetic (PK) profile, and pharmacodynamic (PD) effects on GSBR-1290 in healthy overweight/obese volunteers (HOV) and Type 2 Diabetes Mellitus on Metformin (T2DM) This study includes 5 planned cohorts. Participants will receive multiple-ascending doses of GSBR-1290 or Placebo from Day 1 to Day 84

ELIGIBILITY:
Inclusion Criteria cohorts 1-4:

1. Provided evidence of a signed consent
2. Age ≥ 18 and ≤ 75 years
3. Healthy overweight/obese adult men and women with body mass index ≥ 27 and ≤ 40 kg/m2
4. No nicotine use
5. Have a suitable venous access for blood sampling

Inclusion Criteria cohort 5:

1. Men and women with T2DM of ≥6 months duration
2. Age ≥ 18 and ≤ 75 years
3. BMI ≥ 27 and ≤ 40 kg/m2
4. Treated with stable doses of ≥500 mg of metformin with a duration ≥6 months and at stable doses for ≥2 months with a screening HbA1c ≥7.0% and ≤10.5%.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or major surgery within the major 3 months
2. A sitting BP after resting for 5 minutes > 160mm Hg systolic or > 100 mm Hg diastolic or an apical pulse rate <50 or >100 beats per minute.
3. Evidence of abnormality on the screening visit ECG, or a history of known arrhythmia or prolonged QTcF pr prolonged QRS interval
4. Liver function test results elevated > 2.0-fold above the ULN for gamma glutamyl transferase, alkaline phosphatase, aspartate aminotransferase or alanine aminotransferase. Bilirubin above the ULN
5. Estimated glomerular filtration rate < 60mL/min/1.73 m2 body surface area
6. Known hypersensitivity to any of the study drug ingredients
7. Any other condition or prior therapy that would make the participant unsuitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and relationship of AE/SAE, vital signs, laboratory measures and ECG to assess safety and tolerability of multiple oral doses of GSBR-1290 in HOV and T2DM | 42 days

SECONDARY OUTCOMES:
Analysis of Cmax at specified timepoints predose and postdose to calculate PK parameters | 31 days
Analysis of Tmax at specified timepoints predose and postdose to calculate PK parameters | 31 days
Analysis of AUC at specified timepoints predose and postdose to calculate PK parameters | 31 days
Identification of GSBR-1290 metabolites following oral administration of multiple doses in plasma | 31 days

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, Anaheim, California
  - ProSciento, Inc, Chula Vista, California
  - QPS Miami Research Associates, Miami, Florida
  - Progressive Medical Research, Port Orange, Florida

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol
Time Frame: Data sharing requests will be considered beginning 36 months after the study publication (manuscript accepted for publication) and either 1) the product have been granted marketing authorization in at least two regulatory jurisdictions, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Researchers will submit a request containing the research objectives, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). Structure Therapeutics does not grant external requests for individual de-identified patient data for the following purposes:
  * re-evaluating safety and efficacy end points already addressed in the product labelling,
  * assessing safety or efficacy for an indication in current development
  Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a panel of external advisors. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement.